CLINICAL TRIAL: NCT00534768
Title: Postoperative Treatment After Endoscopic Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH5551813
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Last update posted 2008-01-14 (Estimated); Status verified 2008-01

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis | interventions — Control Groups

ARMS (2):
- 1 (Active Comparator): debridement on 1st, 3-5th and 7th postoperative days
  Interventions: Procedure: active debridement
- 2 (Active Comparator)
  Interventions: Procedure: control group

INTERVENTIONS:
Procedure: active debridement — debridement on 1st, 3-5th and 7th postoperative days
  Arms: 1
Procedure: control group — Postoperative debridement on 7th postoperative day
  Arms: 2

SUMMARY:
Objective: Even though postoperative debridement is commonly considered as an essential part of endoscopic sinus surgery (ESS), the scientific data on the efficacy or the optimal timing of debridement is limited. In the present study, the effect of repeated debridement during the first week after ESS on the endoscopic and subjective outcome was evaluated.

Study Design: Open, prospective, randomized, controlled clinical trial with two parallel groups.

Methods: A total of 90 patients suffering from either recurrent or chronic maxillary sinusitis were randomized into two groups after ESS. In the active group, the nasal cavities were debrided three times on the first postoperative week, while in the control group the patients were debrided only once on the 7th postoperative day. The primary outcome measure was the presence of scarring in the middle meatus at four weeks after ESS.

ELIGIBILITY:
Inclusion Criteria:

* A total of 90 patients (age 18-70 years), who underwent ESS in Kuopio University Hospital, Kuopio, Finland were included in this study.
* The patients suffered from either recurrent or chronic maxillary sinusitis and had American Society of Anaesthesiologists physical status 1 or 2.{{331 Sakland,M. 1941; }}

Exclusion Criteria:

The patients were excluded if they had:

* Undergone previous sinus surgery or if they had severe nasal polyposis (radiological opacification more than 50 % of the sinuses (Lund-McKay classification)
* Hemorrhagic diathesis
* Liver or kidney dysfunction
* Chronic malnutrition
* Alcoholism or inflammatory bowel disease.

Other exclusion criteria were pregnancy and ongoing anticoagulant therapy.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2003-01

PRIMARY OUTCOMES:
scarring in middle meatus 4 weeks after ESS | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tatu p Kemppainen, MD, Principal Investigator — Kuopio University Hospital; Juhani Nuutinen, PhD, Study Director — Kuopio University
Locations (1):
- Kuopio University Hospital, Kuopio, Finland